CLINICAL TRIAL: NCT00676351
Title: Follow up of Ventilatory Function in Infant After One (or More) Bronchiolitis During the First Year of Life. Course Towards Asthma
Brief Title: Follow up of Ventilatory Function in Infant After Bronchiolitis During the First Year of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Cynthia GIRAN, Département de la recherche Clinique et de l'Innovation - CHU de Nice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02-PHRC-05
Record Dates: First submitted 2008-05-12; First posted 2008-05-13 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2008-05

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): body plethysmography Same tests were performed at 18 and 24 months. At 30 and 36 months, pulmonary function was evaluated by measuring respiratory resistances using an oscillometry system and an occlusion system
  Interventions: Procedure: body plethysmography

INTERVENTIONS:
Procedure: body plethysmography — Same tests were performed at 18 and 24 months. At 30 and 36 months, pulmonary function was evaluated by measuring respiratory resistances using an oscillometry system and an occlusion system

SUMMARY:
A significant proportion of asthma is diagnosed during childhood. Bronchiolitis is the most common lower respiratory tract illness (LRI) in early life and the present work is a prospective study undertaken to highlight the possible relationship between LRI in early life and trigger of atopy and asthma in 3 year-old childhood, using paediatric lung function testing.

Twenty nine infants (8 females and 21 males) were included in our study. The beginning of the study started at least three weeks after the first bronchiolitis episode. Pulmonary function test was realized using an infant specific body plethysmography (Babybody, Erich Jaeger, Germany). Same tests were performed at 18 and 24 months. At 30 and 36 months, pulmonary function was evaluated by measuring respiratory resistances using oscillometry and occlusion systems (Masterlab-IOS, Erich Jaeger, Germany). If measured data showed an obstruction, a bronchodilatator was inhaled to assess reversibility. When results were normal, a bronchial provocation test, using inhaled metacholine, was performed.

Skin prick tests (SPTs) were performed during the first exam, and at 24 and 36 months (Stallergenes-DHS).

Collection of data was largely incomplete due to a number of patients lost of follow up. Based on the available data, it can be conclude that most of lung tests results were in the normal range but a non negligible bronchial hyper reactivity was documented (41% of patients).

This study must be continued to increase the number of included patients and to continue their follow up during a longer time.

DETAILED DESCRIPTION:
Asthma affects a large population throughout the world and about two millions of persons in France, killing two hundred patients by year. A significant proportion of cases of asthma are diagnosed during childhood. Understanding the relation between early-life infectious exposures and asthma and atopy appears to be considerable interest.

Respiratory infectious illnesses, mostly viral, are very common in childhood. Bronchiolitis is the most common lower respiratory tract illness (LRI) in early life (1). It is commonly caused by respiratory syncytial virus (RSV) and is often associated with subsequent wheezing and childhood asthma (2). Respiratory infectious illnesses caused by other agent than RSV can be also associated with asthma and atopy (3). However, the relation between respiratory infectious illnesses in early life and asthma in childhood is again much debated since some studies show a relationship between bronchiolitis and atopy (4) but not others (5, 6).

The present work is a prospective study undertaken to highlight the possible relationship between LRI in early life and trigger of atopy and asthma in 3 year-old childhood, using paediatric lung function testing.

Twenty nine infants (8 females and 21 males) were included in our study and 8 of 29 infants were of premature birth. The youngest patient was 3 months old and the older fourteen months old. The beginning of the study started at least three weeks after the first bronchiolitis episode. Pulmonary function test was realized using body plethysmography (Babybody, Erich Jaeger, Germany). Same tests were performed at 18 and 24 months. At 30 and 36 months, pulmonary function was evaluated by measuring respiratory resistances using an oscillometry system and an occlusion system (Masterlab-IOS, Erich Jaeger, Germany). All respiratory tests were performed on patients in asymptomatic respiratory condition and at least one month apart from respiratory infection. If measured data showed an obstruction, a bronchodilator was inhaled to assess reversibility. When results were normal, a bronchial provocation test, using inhaled metacholine, was performed.

Skin prick tests (SPTs) were performed at the first exam, and at 24 and 36 months (Stallergenes-DHS). Dermatophagoides pteronyssinus, alternaria, cat dander, cockroach, orchard grass and timothy grass were systematically tested. The SPTs were considered positive when the wheal diameter was over 3 mm and 50% larger than the positive control, and the negative control remained negative (7). The possibility of dermographism was eliminated by a negative reaction of the negative control.

Collection of data was largely incomplete due to a number of patients lost of follow up. Briefly, based on the available data, most of lung tests results were in the normal range although a proportion of patients experienced recurrent wheezing episodes during follow up. Nevertheless a bronchial hyper reactivity to metacholine was documented in 41%. Atopy, as screened by SPTs, was detected in a minority of infants (13.5%). Coexistence of bronchial hyper reactivity and atopy was present in only one patient.

These incomplete results highlight the complex interplay between symptoms, bronchial obstruction, bronchial hyper reactivity and atopy in the subsequent development of asthma in wheezy children. Long term follow up is necessary to assess the prognostic value of these parameters.

ELIGIBILITY:
Inclusion Criteria:

* child under 32 months old
* child suffering from bronchiolitis episode at least 3 weeks before beginning the study

Exclusion Criteria:

* child over 32 months old
* child suffering from bronchiolitis episode since less than 3 weeks

Ages: 3 Months to 32 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2004-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Body plethysmography at least three weeks after the first bronchiolitis episode and at 18 and 24 months | 18, 24, 30 and 36 months
Respiratory resistances measure (oscillometry and occlusion systems) at 30 and 36 months | 18, 24, 30 and 36 months

SECONDARY OUTCOMES:
Skin prick tests | at the first exam, and at 24 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique CRENESSE, PU PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CRENESSE Dominique, Nice, France

REFERENCES:
- [Background] Wright AL, Taussig LM, Ray CG, Harrison HR, Holberg CJ. The Tucson Children's Respiratory Study. II. Lower respiratory tract illness in the first year of life. Am J Epidemiol. 1989 Jun;129(6):1232-46. doi: 10.1093/oxfordjournals.aje.a115243. PMID 2729259
- [Background] Sigurs N, Gustafsson PM, Bjarnason R, Lundberg F, Schmidt S, Sigurbergsson F, Kjellman B. Severe respiratory syncytial virus bronchiolitis in infancy and asthma and allergy at age 13. Am J Respir Crit Care Med. 2005 Jan 15;171(2):137-41. doi: 10.1164/rccm.200406-730OC. Epub 2004 Oct 29. PMID 15516534
- [Background] Van Bever HP, Wieringa MH, Weyler JJ, Nelen VJ, Fortuin M, Vermeire PA. Croup and recurrent croup: their association with asthma and allergy. An epidemiological study on 5-8-year-old children. Eur J Pediatr. 1999 Mar;158(3):253-7. doi: 10.1007/s004310051062. PMID 10094451
- [Background] Schauer U, Hoffjan S, Bittscheidt J, Kochling A, Hemmis S, Bongartz S, Stephan V. RSV bronchiolitis and risk of wheeze and allergic sensitisation in the first year of life. Eur Respir J. 2002 Nov;20(5):1277-83. doi: 10.1183/09031936.02.00019902. PMID 12449185
- [Background] Stein RT, Sherrill D, Morgan WJ, Holberg CJ, Halonen M, Taussig LM, Wright AL, Martinez FD. Respiratory syncytial virus in early life and risk of wheeze and allergy by age 13 years. Lancet. 1999 Aug 14;354(9178):541-5. doi: 10.1016/S0140-6736(98)10321-5. PMID 10470697
- [Background] Sampson HA, Albergo R. Comparison of results of skin tests, RAST, and double-blind, placebo-controlled food challenges in children with atopic dermatitis. J Allergy Clin Immunol. 1984 Jul;74(1):26-33. doi: 10.1016/0091-6749(84)90083-6. PMID 6547461